CLINICAL TRIAL: NCT07280377
Title: A Phase 1 / 2 Multiple-indication Biomarker, Safety, and Efficacy Study in Advanced or Metastatic Gastrointestinal Cancers Exploring Treatment Combinations With Pelareorep and Atezolizumab
Brief Title: A Study in Advanced or Metastatic Gastrointestinal Cancers Exploring Treatment Combinations With Pelareorep and Atezolizumab
Acronym: GOBLET
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oncolytics Biotech (Industry)
Collaborators: Crolll Gmbh (Other); AIO-Studien-gGmbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REO 029; 2024-515936-62-00 (EU CTIS Number); 2020-003996-16 (EudraCT Number)
Record Dates: First submitted 2025-11-18; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Anal Cancer Metastatic; Squamous Cell Carcinoma of the Anus Stage Unspecified; Pancreatic Cancer Metastatic; Unresectable Pancreatic Carcinoma
MeSH Terms: interventions — reolysin; atezolizumab; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: Metastatic Pancreatic Cancer 1L (Experimental): Patients with first-line (1L) locally advanced/metastatic unresectable pancreatic ductal adenocarcinoma (PDAC): Pelareorep and atezolizumab added to gemcitabine and nab-paclitaxel
  Interventions: Drug: Pelareorep; Drug: Atezolizumab; Drug: Gemcitabine and nab-paclitaxel
- Cohort 2: Metastatic Colorectal Cancer 1L (MSI-H/dMMR) (Experimental): Patients with 1L metastatic colorectal cancer (mCRC), limited to microsatellite instability-high (MSIH) or mismatch repair deficient (dMMR) tumors: Pelareorep and atezolizumab
  Interventions: Drug: Pelareorep; Drug: Atezolizumab
- Cohort 3: Metastatic Colorectal Cancer 3L (Experimental): Patients with third-line (3L) mCRC independent of microsatellite instability (MSI)/dMMR status: Pelareorep and atezolizumab added to trifluridine/tipiracil
  Interventions: Drug: Pelareorep; Drug: Atezolizumab; Drug: Trifluridine Tipiracil
- Cohort 4: Metastatic Unresectable Anal Cancer >/=2L (Experimental): Patients with >/= 2L locally advanced/metastatic unresectable squamous cell carcinoma of the anal canal (SCCA) of viral or non-viral origin after prior systemic chemotherapy: Pelareorep and atezolizumab
  Interventions: Drug: Pelareorep; Drug: Atezolizumab
- Cohort 5: Metastatic PDAC 1L (Experimental): Patients with 1L metastatic PDAC: Pelareorep and modified FOLFIRINOX (mFOLFIRINOX) with or without atezolizumab
  Interventions: Drug: Pelareorep; Drug: Atezolizumab; Drug: mFOLFIRINOX Treatment Regimen

INTERVENTIONS:
Drug: Pelareorep — Pelareorep 4.5 x 10^10 TCID50 via 1-hour IV infusion
Drug: Atezolizumab — Atezolizumab 840 mg IV infusion
  Other Names: Tecentriq
Drug: Gemcitabine and nab-paclitaxel — Gemcitabine (1,000 mg/m2) and nab-paclitaxel (125 mg/m2)
  Other Names: Gemzar; Abraxane
  Arms: Cohort 1: Metastatic Pancreatic Cancer 1L
Drug: Trifluridine Tipiracil — Trifluridine/tipiracil administered at a 35 mg/m2 dose orally twice daily
  Other Names: Lonsurf
  Arms: Cohort 3: Metastatic Colorectal Cancer 3L
Drug: mFOLFIRINOX Treatment Regimen — mFOLFIRINOX- IV oxaliplatin 85 mg/m2; IV leucovorin 400 mg/m2; IV irinotecan 150 mg/m2; 5-FU 2400 mg/m2 by 46-hour infusion, per local standard of care
  Arms: Cohort 5: Metastatic PDAC 1L

SUMMARY:
This is an open-label, phase 1/2, multiple-indication platform study to explore safety, potential predictive immune-related biomarkers, and early efficacy (as measured by objective response rate [ORR; Cohorts 1,2, 4,and 5] and disease control rate [DCR; Cohort 3]) in patients with advanced or metastatic gastrointestinal (GI) tumors. Cohorts 1-4 are not randomized; however, Cohort 5 is comprised of two treatment arms to which patients are randomized in a 1:1 ratio.

DETAILED DESCRIPTION:
The overall aim is to assess safety, predictive biomarkers, and preliminary efficacy as assessed by tumor response criteria at week 16 for cohorts1, 2, 3, and 4, and best overall response rate and OS in Cohort 5. If a cohort shows a promising ORR in Stage 1 of the Simon two-stage design, that cohort may be expanded to enroll additional patients (up to 50 patients in Cohorts 1 and 3 , up to 28 patients in Cohort 4, and up to 64 patients in Cohort 5) in an extension phase per predetermined statistical conditions. In addition, either or both arms of Cohort 5 may expand if the data collected in Stage 1 suggest that expansion may help in assessing the potential survival benefit of the investigational therapy(ies). In this study, we hypothesize that treatment with pelareorep will prime the tumor microenvironment (TME) for checkpoint blockade therapy, thereby increasing PD-L1 expression and the number of new T cell clones within the tumor, both of which are associated with increased response to checkpoint blockade.

ELIGIBILITY:
Cohorts 1-5 Inclusion Criteria:

* ECOG performance status of 0 or 1
* Have measurable lesions per RECIST v1.1
* Patients must have adequate hematological, renal, and hepatic function
* Have recovered to ≤grade 1 or baseline for all adverse events (AEs) due to previous therapies or surgeries.
* For female patients of childbearing potential and male patients with partners of childbearing potential, agreement to use a highly-effective form(s) of contraception and to continue its use for 6 months after the last dose of study drug.

Exclusion Criteria:

* Undergone systemic chemotherapy, radiotherapy, or surgery, <4 weeks before study treatment.
* Received previous treatment with immune checkpoint inhibitors
* Uncontrolled or severe cardiac disease
* Active, uncontrolled infections
* Symptomatic brain metastasis
* Interstitial lung disease with symptoms or signs of activity.
* Autoimmune disease that has required systemic treatment in the past 2 years with disease modifying agents, corticosteroids, or immunosuppressive drugs.
* A seizure disorder that requires pharmacotherapy.
* Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation.
* A non-healing wound, non-healing ulcer, or non-healing bone fracture within 4 weeks prior to the start of study drug.
* Women who are pregnant or breastfeeding.
* A diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy
* Any vaccine within 28 days prior to first treatment or during the first cycle of study treatment.

Exclusion Criteria:

* In Cohort 1, 2, 3, 4: Life expectancy less than 3 months
* In Cohort 1, 2, 3: known active Hepatitis B (HBV) or Hepatitis C (HCV) infection that requires anti-viral treatment.
* In Cohort 4: Prior HIV infection if the CD4+ T cell is <300 cells/µl
* In Cohort 5: Known low or absent dihydropyrimidine dehydrogenase (DPD) activity.
* In Cohort 5: Known leptomeningeal disease.
* In Cohort 5: History of another primary cancer within the last 3 years with the exception of non-melanoma skin cancer, early-stage prostate cancer, or curatively treated cervical carcinoma in-situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) for Cohort 1, 2, 4, and 5 | At week 16 (within each cohort)
  Proportion of patients with complete response [CR], partial response [PR] assessed by the investigators and/or central reader according to RECIST v1.1
Disease Control Rate (DCR) - Cohort 3 | at week 16
  DCR (complete response [CR], partial response [PR], and stable disease [SD]) assessed by the investigators according to RECIST v 1.1.
Overall Survival (OS) - Cohort 5 | Cohort 5: From the date of randomization through long term follow up at 2 years
  OS is defined as the time from date of first treatment to death from any cause

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From initiation of treatment to objective progression or death from any cause, whichever occurs first, up to two years
  Time from the first dose date of study treatment to the date of investigator-determined objective progression (according to RECIST 1.1) or death from any cause, whichever occurs first.
Duration of Response (DOR) | From initiation of treatment to disease progression or death from any cause, whichever occurs first, up to two years
  Time from documentation of the first CR or PR to the time of first documented evidence of progressive disease (or relapse for subjects who experience CR during the study) or death.
Disease Control Rate (DCR) | From initiation of treatment to disease progression or death from any cause, whichever occurs first, up to two years
  Overall DCR, defined as the number of patients with a best overall response of CR, PR, or SD according to RECIST v. 1.1.
Overall Response Rate (ORR) - Cohort 1-4 | From initiation of treatment to disease progression or death from any cause, whichever occurs first, up to two years
  ORR, defined as the percentage of patients with a best overall response of complete response [CR] or partial response [PR] according to RECIST v 1.1, and confirmed ORR, defined as the percentage of patients with a CR or PR at two or more consecutive evaluation timepoints.
Overall Survival (OS) - Cohort 1-4 | From the date of randomization through long term follow up at 3 years
  OS defined as the time from date of first treatment to death from any cause

CONTACTS AND LOCATIONS:
Locations (15):
- Germany (15):
  - Nationales Centrum für Tumorerkrankungen Heidelberg, Heidelberg, Baden-Wurttemberg
  - SLK-Kliniken Heilbronn GmbH, Heilbronn, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Gemeinschaftspraxis Dr. Med Bernhard Heinreich, Augsburg, Bavaria
  - Klinikum der Universität München, München, Bavaria
  - Hämatologisch-Onkologische Praxis Eppendorf, Hamburg, Hamburg
  - Asklepios Kliniken Hamburg GmbH, Hamburg, Hamburg
  - Krankenhaus Nordwest, Frankfurt am Main, Hesse
  - St. Josef-Hospìtal, Bochum, Bochum, North Rhine-Westphalia
  - Universitätsmedizin Mainz, Mainz, Rhineland-Palatinate
  - Caritasklinikum Saarbrücken St. Theresia, Saarbrücken, Saarland
  - Klinikum Chemnitz gGmbH, Chemnitz, Saxony
  - Universität Leipzig, Leipzig, Saxony
  - Charité Universitätsklinikum Berlin, Berlin, State of Berlin